## **Study Informed Consent Form**

# HEmodynamic Resuscitation and Monitoring in Early Sepsis (HERMES Study)

# An ISCCM research project



### **Principle Investigator:**

Prof. Sheila Nainan Myatra Tata Memorial Hospital, Mumbai, INDIA

Email: sheila150@hotmail.com Cell: 9820156070

# Short consent of Legally acceptable representative for HERMES study Title-: Hemodynamic Resuscitation and Monitoring in Early Sepsis (HERMES Study)

I understand that a study "Hemodynamic Resuscitation and Monitoring in Early Sepsis (HERMES Study)." conducted by Dr. Sheila Nainan Myatra Professor, Department of Anesthesiology, Critical Care and Pain, Tata Memorial Hospital, Parel, Mumbai Mob No 9820156070" involves the analysis of my relatives medical data that has been collected as part of my routine medical care.

I understand that the principal investigator is conducting this study to capture the patient characteristics, practices regarding treatment and observation measures required to maintain the blood pressure in patient presenting with early infection and low blood pressure to Indian ICUs. I also understand that principal investigator is also trying to find out the various factors associated with improved survival in patients with low blood pressure caused by infection.

I also understand that there will not be any additional medical procedures over and above those which my patient will encounter during standard treatment. I also understand this study only involved data collection regarding to resuscitation practices that my patient is receiving as a part of his routine medical care.

I understand that this study has been approved by the Institutional Ethics Committee, Tata Memorial Centre and does not pose any additional risk to my relative beyond that which my patient will encounter while undergoing routine physical or psychological examinations or tests and/or which my patient would encounter in routine daily life activities. I further understand that confidentiality with regard to my relative's medical data will be ensured, and that the results published will not in any way be linked to my relative. I understand that the Principal Investigator Dr. Sheila Nainan Myatra will be willing to provide me with any additional information that I would want to know regarding the study.

I understand that if I decline to participate in this study or withdraw my consent at any stage of the study my relative's medical treatment will not be affected.

If you have any queries at any time about the study or the procedures, or you experience adverse effect as a result of participating in this study, you may contact,

### Dr. Sheila N Myatra, Professor,

Department of Anesthesiology, Critical Care and Pain, Tata Memorial Hospital, Parel, Mumbai – 400 012, Tel: 9820156070, Email- sheila150@hotmail.com

If you have questions about your rights as a participant, then contact the,

Dr. Umesh Mahantshetty (IEC-I)/ Dr. Girish Chinnasamy (IEC-II)

Member Secretary, Institutional Ethics Committee

Tata Memorial Hospital,

Dr E. Borges Rd., Mumbai-400012 Tel no- 022 24177262

Participant's name: Legal Acceptable Representative name Legal Acceptable Representative signature/Thumb Impression & date (if applicable): Impartial Witness's name: Impartial Witness's signature & date (if applicable): Name of PI or Co-PI/Co-I: PI or Co-PI/Co-I sign & date:

I am willing to allow the use of my/ my relative's data for the study.